CLINICAL TRIAL: NCT01372020
Title: The Effect of Neuromuscular Electrical Therapy on Pain in Patients With Venous Ulcers: a Controlled Clinical Trial
Brief Title: Neuromuscular Electrical Therapy in Venous Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Faculdade Evangelica do Parana (Other)
Responsible Party: Principal Investigator, Silvia Valderramas, Silvia Valderramas, Faculdade Evangelica do Parana
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fepar-04
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Venous Insufficiency
Keywords: Varicose ulcer; wound healing; electrical stimulation
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Sham Comparator)
  Interventions: Other: neuromuscular electrical stimulation
- neuromuscular electrical therapy (Experimental)
  Interventions: Other: neuromuscular electrical stimulation

INTERVENTIONS:
Other: neuromuscular electrical stimulation — The application technique used will be bipolar, with electrodes of the type metal-tipped pen. The electrodes will be placed at the outer edges of the ulcer, on opposite sides of the same and the estimated time of 1 minute at each point. All the edge of the ulcer will be bypassed, thereby separating the injections every 1 cm, returning to the starting point at the end of the application. To ensure that the entire edge of the ulcer to receive the stimulation, the end points of the application, the application will be made for another minute sliding the pen around the whole edge. Thus the application time will be directly proportional to the ulcer area. The subjects will be received 10 applications, three times a week for a period of 4 weeks.
  Other Names: intervention group

SUMMARY:
The use of neuromuscular electrical stimulation in the treatment of venous ulcers with difficulty of repair could be an alternative therapeutic favoring devitalized tissues and hence the pain.

The aim of this study is to evaluate the effect of neuromuscular electrical stimulation on pain and area of venous ulcers in patients with venous insufficiency.

DETAILED DESCRIPTION:
The aim was to evaluate the effect of neuromuscular electrical stimulation on pain and area of venous ulcers in patients with venous insufficiency. In a simple-blind controlled clinical study, 20 subjects with venous ulcers with age over 50 years will be divided in two groups:neuromuscular electrical stimulation(n=10) and control group (n=10). Pain (by Visual Analogue Scale) and the ulcer area (by planimetry on graph paper and the software ImageJ ®) were measured.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders
* aged over 50 years
* sedentary and with clinical diagnosis of chronic venous insufficiency with ulcer in lower limbs will be included

Exclusion Criteria:

* Subjects with pacemakers
* diabetes
* uncontrolled hypertension
* osteomyelitis and pain of unknown origin
* unable to walk or make use of drugs that acted directly on the healing process will be excluded

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pain | the subjects will be followed for a period of 4 weeks.
  Pain assessment will be performed by the Visual Analogue Scale

SECONDARY OUTCOMES:
ulcer area | the patients will be folloed for the 4-weeks.
  the ulcer area will be measured by the planimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Korelo Raciele, M.sC, Principal Investigator — Facukdade Dom Bosco
Locations (1):
- Faculdade Dom Bosco, Curitiba, Paraná, Brazil

REFERENCES:
- [Result] Carley PJ, Wainapel SF. Electrotherapy for acceleration of wound healing: low intensity direct current. Arch Phys Med Rehabil. 1985 Jul;66(7):443-6. PMID 3893385
- [Derived] Korelo RI, Valderramas S, Ternoski B, Medeiros DS, Andres LF, Adolph SM. Microcurrent application as analgesic treatment in venous ulcers: a pilot study. Rev Lat Am Enfermagem. 2012 Jul-Aug;20(4):753-60. doi: 10.1590/s0104-11692012000400016. English, Portuguese, Spanish. PMID 22990161